CLINICAL TRIAL: NCT00548925
Title: A Global, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of ABT-894 Versus Placebo in Subjects With Diabetic Neuropathic Pain
Brief Title: A Safety and Efficacy Study in Subjects With Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-014; 2007-001140-47 (EudraCT Number)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuropathic Pain
MeSH Terms: interventions — 3-(5,6-dichloropyridin-3-yl)-3,6-diazabicyclo(3.2.0)heptane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ABT-894
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-894 — 6 mg BID tablets, 8 weeks of treatment
  Arms: 1
Drug: placebo — BID tablets, 8 weeks of treatment
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a 6 mg twice a day dose of an investigational product in subjects with diabetic neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 75
* If female, must be of non-childbearing potential or practicing birth control
* Has diabetes mellitus (Type 1 or 2) and a diagnosis of painful distal symmetric diabetic polyneuropathy
* Has had pain from distal symmetric diabetic polyneuropathy for a minimum of 6 months
* Must be willing to washout of all analgesic medications prior to entry into the study

Exclusion Criteria:

* Has other conditions that may cause pain
* Currently receiving analgesic medications for conditions other than diabetic neuropathic pain
* Has a history of certain psychiatric diseases
* Has a history of certain heart or cardiovascular conditions
* Has any clinically significant recent infection, injury, or illness
* Current participation in another clinical study or participation within the past 30 days
* Is incapacitated, bedridden or confined to a wheelchair
* Is pregnant and/or breastfeeding
* Previous participation in this study or any other study with this investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Weekly mean of 24-hour average pain score | Change from Baseline to final

SECONDARY OUTCOMES:
Pain improvement from Baseline to the final evaluation | 8-week
Weekly mean of 24-hour worst pain severity; weekly average night pain and morning pain | 8-week
Global assessments of study drug and pain status | 8-week
Short-Form McGill Pain Questionnaire (SF-MPQ), Neuropathic Pain Scale (NPS) | 8-week

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Duan, MD, Study Director — AbbVie
Locations (29):
- United States (12):
  - Site Reference ID/Investigator# 6614, Spring Valley, California
  - Site Reference ID/Investigator# 6617, Walnut Creek, California
  - Site Reference ID/Investigator# 6356, Hollywood, Florida
  - Site Reference ID/Investigator# 6615, Tampa, Florida
  - Site Reference ID/Investigator# 6358, Wellington, Florida
  - Site Reference ID/Investigator# 6609, St Louis, Missouri
  - Site Reference ID/Investigator# 7229, New Hyde Park, New York
  - Site Reference ID/Investigator# 6618, Charlotte, North Carolina
  - Site Reference ID/Investigator# 6607, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 6575, Allentown, Pennsylvania
  - Site Reference ID/Investigator# 8179, San Antonio, Texas
  - Site Reference ID/Investigator# 6616, San Antonio, Texas
- Czechia (3):
  - Site Reference ID/Investigator# 5552, Hradec Králové
  - Site Reference ID/Investigator# 5554, Olomouc
  - Site Reference ID/Investigator# 5553, Zlín
- France (3):
  - Site Reference ID/Investigator# 9363, Corbeil-Essonnes
  - Site Reference ID/Investigator# 5557, Limoges
  - Site Reference ID/Investigator# 6238, Nevers
- Germany (5):
  - Site Reference ID/Investigator# 6564, Bad Mergentheim
  - Site Reference ID/Investigator# 11201, Berlin
  - Site Reference ID/Investigator# 6234, Düsseldorf
  - Site Reference ID/Investigator# 11202, Mainz
  - Site Reference ID/Investigator# 7714, Munich
- Italy (2):
  - Site Reference ID/Investigator# 5549, L’Aquila
  - Site Reference ID/Investigator# 5558, Perugia
- Spain (2):
  - Site Reference ID/Investigator# 6475, Granada
  - Site Reference ID/Investigator# 7911, Sabadell, Barcelona
- United Kingdom (2):
  - Site Reference ID/Investigator# 5555, Birmingham
  - Site Reference ID/Investigator# 7133, Sheffield